CLINICAL TRIAL: NCT06232018
Title: A Comparison of 2-octyl Cyanoacrylate Skin Adhesive and Polyester Mesh for Wound Closure in Total Knee Arthroplasty, A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pooriwat Lertsurawat (Other)
Collaborators: Kittipon Naratrikun (Unknown)
Responsible Party: Sponsor-Investigator, Pooriwat Lertsurawat, Resident Orthopedic of Hatyai Hospital, HatYai Hospital
Organization: HatYai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HYH EC 059-66-01
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: OsteoArthritis Knee
Keywords: Dermabond; Dermabond prineo
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Skin adhesive (Experimental): 2-octylcyanoacrylate glue (DERMABOND ADVANCED®, Ethicon, johnson & johnson, Somerville, NJ)
  Interventions: Device: Skin adhesive (Dermabond)
- skin adhesive Plus polyester mesh (Active Comparator): 2-octylcyanoacrylate glue + polyester mesh ( DERMABOND PRINEO®, Ethicon, johnson & johnson, Somerville, NJ)
  Interventions: Device: skin adhesive + polyester mesh (Dermabond prineo)

INTERVENTIONS:
Device: Skin adhesive (Dermabond) — * Arthrotomy (deep layer) is repaired using number 1-0 monofilament absorbable suture (STRATAFIX™ , Ethicon, johnson & johnson, Somerville, NJ)
  * Subcuticular suture is repaired using number 3-0 monofilament absorbable suture (STRATAFIX™ , Ethicon, johnson & johnson, Somerville, NJ)
  * After subticular sutures was done
  * 2-octylcyanoacrylate glue (DERMABOND ADVANCED®, Ethicon, johnson & johnson, Somerville, NJ) was applied
  Arms: Skin adhesive
Device: skin adhesive + polyester mesh (Dermabond prineo) — * Arthrotomy (deep layer) is repaired using number 1-0 monofilament absorbable suture (STRATAFIX™ , Ethicon, johnson & johnson, Somerville, NJ)
  * Subcuticular suture is repaired using number 3-0 monofilament absorbable suture (STRATAFIX™ , Ethicon, johnson & johnson, Somerville, NJ)
  * After subticular sutures was done
  * 2-octylcyanoacrylate glue + polyester mesh ( DERMABOND PRINEO®, Ethicon, johnson & johnson, Somerville, NJ) was applied
  Arms: skin adhesive Plus polyester mesh

SUMMARY:
The goal of this randomized controlled study is to investigate the Efficacy of Using skin adhesive (Dermabond) and skin adhesive with polyester mesh (Dermabond Prineo )for Wound Closure in Total Knee Arthroplasty, The main question it aim to answer

1 Are skin adhesive alone and with Polyester mesh in Total knee arthroplasty different in Patient satisfaction evaluated by POSAS score

DETAILED DESCRIPTION:
Nowadays, there are many methods of wound closure in Total Knee arthroplasty, such as nylon, skin staple, and sterile strip, which differ in advantages and disadvantages of each technique. However, these methods have the same disadvantages: wound discharge, which may lead to infection, wound separation, and the need for wound dressing. It is also a burden for patients and caregivers. In travelling to change the wound in a hospital, There are many costs in terms of wound dressing equipment, travel costs and time off from work for caregivers to take patients to get wound dressing.

Skin adhesive is an innovation for wound closure in total knee arthroplasty. It reduces the problem of wound separation, with no need for wound dressing.

Skin adhesive mesh has been studied in many studies, showing that it can be used well. Strong It is no different from traditional wound closure; the scar is more beautiful. Patients are more satisfied. But the disadvantage is the high price.

Skin adhesive without polyester mesh has the advantage of being cheaper three times than polyester mesh but less intense than with mesh. This makes it unpopular.

No studies have been found comparing wound dressings with mesh and no mesh After knee replacement surgery.

Therefore, this study is to compare skin adhesive and skin adhesive plus polyester mesh in closure wound total knee arthroplasty.

Are there differences in patient satisfaction Are wound complications such as wound oozing, wound separation, superficial wound skin infection, and contact dermatitis different?

ELIGIBILITY:
Inclusion Criteria:

* OA knee need for Total knee arthroplasty
* Age 50-80 years old

Exclusion Criteria:

* Previous surgery of knee
* History of Keloid, Scar, Psoriasis at the knee
* History of contact dermatitis with skin adhesive
* Cognitive impairment

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pooriwat Lertsurawat, Songkhla, Changwat Songkhla, Thailand

REFERENCES:
- [Background] Kong X, Yang M, Guo R, Chen J, Chai W, Wang Y. A Prospective, Randomized and Controlled Study on Tissue Adhesive for Skin Incision in Total Knee Arthroplasty. Ther Clin Risk Manag. 2020 Aug 24;16:795-802. doi: 10.2147/TCRM.S260007. eCollection 2020. PMID 32922017
- [Background] Sundaram K, Piuzzi NS, Patterson BM, Stearns KL, Krebs VE, Mont MA. Skin closure with 2-octyl cyanoacrylate and polyester mesh after primary total knee arthroplasty offers superior cosmetic outcomes and patient satisfaction compared to staples: a prospective trial. Eur J Orthop Surg Traumatol. 2020 Apr;30(3):447-453. doi: 10.1007/s00590-019-02591-4. Epub 2019 Nov 5. PMID 31691153
- [Background] Choi KY, Koh IJ, Kim MS, Park DC, Sung YG, In Y. 2-Octyl Cyanoacrylate Topical Adhesive as an Alternative to Subcuticular Suture for Skin Closure After Total Knee Arthroplasty: A Randomized Controlled Trial in the Same Patient. J Arthroplasty. 2021 Sep;36(9):3141-3147. doi: 10.1016/j.arth.2021.04.033. Epub 2021 May 3. PMID 34024693
- [Background] Khan RJ, Fick D, Yao F, Tang K, Hurworth M, Nivbrant B, Wood D. A comparison of three methods of wound closure following arthroplasty: a prospective, randomised, controlled trial. J Bone Joint Surg Br. 2006 Feb;88(2):238-42. doi: 10.1302/0301-620X.88B2.16923. PMID 16434531
- [Background] El-Gazzar Y, Smith DC, Kim SJ, Hirsh DM, Blum Y, Cobelli M, Cohen HW. The use of dermabond(R) as an adjunct to wound closure after total knee arthroplasty: examining immediate post-operative wound drainage. J Arthroplasty. 2013 Apr;28(4):553-6. doi: 10.1016/j.arth.2012.07.038. Epub 2012 Oct 29. PMID 23114193
- [Background] Gromov K, Troelsen A, Raaschou S, Sandhold H, Nielsen CS, Kehlet H, Husted H. Tissue Adhesive for Wound Closure Reduces Immediate Postoperative Wound Dressing Changes After Primary TKA: A Randomized Controlled Study in Simultaneous Bilateral TKA. Clin Orthop Relat Res. 2019 Sep;477(9):2032-2038. doi: 10.1097/CORR.0000000000000637. PMID 30811354
- [Background] Kim KY, Anoushiravani AA, Long WJ, Vigdorchik JM, Fernandez-Madrid I, Schwarzkopf R. A Meta-Analysis and Systematic Review Evaluating Skin Closure After Total Knee Arthroplasty-What Is the Best Method? J Arthroplasty. 2017 Sep;32(9):2920-2927. doi: 10.1016/j.arth.2017.04.004. Epub 2017 Apr 12. PMID 28487090

RESULTS

PARTICIPANT FLOW:
Groups:
- Skin Adhesive: 2-octylcyanoacrylate glue (DERMABOND ADVANCED®, Ethicon, johnson & johnson, Somerville, NJ)
  Skin adhesive (Dermabond): - Arthrotomy (deep layer) is repaired using number 1-0 monofilament absorbable suture (STRATAFIX™ , Ethicon, johnson & johnson, Somerville, NJ)
  * Subcuticular suture is repaired using number 3-0 monofilament absorbable suture (STRATAFIX™ , Ethicon, johnson & johnson, Somerville, NJ)
  * After subticular sutures was done
  * 2-octylcyanoacrylate glue (DERMABOND ADVANCED®, Ethicon, johnson & johnson, Somerville, NJ) was applied
- Skin Adhesive Plus Polyester Mesh: 2-octylcyanoacrylate glue + polyester mesh ( DERMABOND PRINEO®, Ethicon, johnson & johnson, Somerville, NJ)
  skin adhesive + polyester mesh (Dermabond prineo): - Arthrotomy (deep layer) is repaired using number 1-0 monofilament absorbable suture (STRATAFIX™ , Ethicon, johnson & johnson, Somerville, NJ)
  * Subcuticular suture is repaired using number 3-0 monofilament absorbable suture (STRATAFIX™ , Ethicon, johnson & johnson, Somerville, NJ)
  * After subticular sutures was done
  * 2-octylcyanoacrylate glue + polyester mesh ( DERMABOND PRINEO®, Ethicon, johnson & johnson, Somerville, NJ) was applied
Period: Overall Study
Arm/Group | Skin Adhesive | Skin Adhesive Plus Polyester Mesh
Started | 40 | 40
Completed | 40 | 38
Not Completed | 0 | 2
Not completed — withdrew due to trauma | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Skin Adhesive | Skin Adhesive Plus Polyester Mesh | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.78 (8.12) | 67.43 (5.97) | 67.61 (6.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 5 | 41
  Male | 4 | 35 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 40 | 40 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: Kg/m2] | 26.89 (3.77) | 28.23 (4.20) | 27.56 (4.02)
Hypertension [Number; unit: participants] | 32 | 34 | 66
Diabetic mellitus [Number; unit: participants] | 6 | 10 | 16
Dyslipidemia [Number; unit: participants] | 27 | 28 | 55
Smoking [Number; unit: participants] | 0 | 1 | 1
Alcohol [Number; unit: participants] | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Patient Observer Scar Assessment Score (POSAS)
Description: Evaluated Patient observer scar assessment score (POSAS)
  * The POSAS is composed of two numerical scales that evaluate signs and symptoms of healing.
  * Consists of the two following parts: a scale for patients and a scale for observers.
  * Both contain six items punctuated numerically from 1 to 10
  * The lowest score is 1 and corresponds to the normal skin
  * The highest score is 10 and corresponds to the worst skin
  * The total score of both scales can be calculated simply by adding the scores of each of the six items.
  * The total score will range from 6 to 60.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Skin Adhesive | Skin Adhesive Plus Polyester Mesh
Number analyzed (Participants) | 40 | 38
score on a scale | 20 (6.56) [14 to 26] | 21 (4.88) [14 to 26]
Statistical Analysis 1: Comparison: Skin Adhesive vs Skin Adhesive Plus Polyester Mesh; The Mann-Whitney U test was used to compare POSAS scores between the two groups at 6 weeks . A two-sided p value < 0.05 was considered statistically significant. The study was powered to detect a mean difference of 5 points in POSAS score with 80% power and a 5% alpha error; Test type: Superiority; p = 0.481, Wilcoxon (Mann-Whitney) — Two-tailed Mann-Whitney U test; significance set at p < 0.05; Median Difference (Final Values) = 1, 95% CI 2-sided [-2 to 4], Standard Deviation 6

2. Secondary Outcome: Patient Observer Scar Assessment Score (POSAS)
Description: as for outcome 1
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Skin Adhesive | Skin Adhesive Plus Polyester Mesh
Number analyzed (Participants) | 40 | 38
score on a scale | 13 [10 to 19] | 15 [10 to 20]
Statistical Analysis 1: Comparison: Skin Adhesive vs Skin Adhesive Plus Polyester Mesh; Test type: Superiority; p = 0.228, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2, 95% CI 2-sided [-1.5 to 5], Standard Deviation 5

3. Secondary Outcome: Vancouver Scar Scale
Description: Evaluated vancouver scar scale
  Vancouver Scar Scale (VSS) is used for validated scar assessment tools. Consist of the four following parts: vascularity(0-3) , height(0-3), pliability(0-5), and pigmentation(0-2). Each characteristic is given a score, which are added together to give an overall score between 0 and 13. The lowest score is 0 and corresponds to the normal skin. The highest score is 13 and corresponds to the worst skin.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: Score (0-13)
Arm/Group | Skin Adhesive | Skin Adhesive Plus Polyester Mesh
Number analyzed (Participants) | 40 | 38
Score (0-13) | 5 [5 to 6] | 5 [5 to 6]
Statistical Analysis 1: Comparison: Skin Adhesive vs Skin Adhesive Plus Polyester Mesh; Test type: Superiority; p = 0.446, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-1 to 1], Standard Deviation 0.5

4. Secondary Outcome: Wound Leakage
Description: Wound leakage was evaluated by measuring the total blood-stained area on the waterproof dressing.
  The dressing was placed on a standardized 1 mm² grid, and the stained area was calculated in square millimeters (mm²).
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: square millimeter (mm²)
Arm/Group | Skin Adhesive | Skin Adhesive Plus Polyester Mesh
Number analyzed (Participants) | 40 | 38
square millimeter (mm²) | 23 [9.8 to 57.5] | 79 [42.8 to 108.8]
Statistical Analysis 1: Comparison: Skin Adhesive vs Skin Adhesive Plus Polyester Mesh; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 56, 95% CI 2-sided [40 to 70], Standard Deviation 25

5. Secondary Outcome: Vancouver Scar Scale
Description: as for outcome 3
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: Score (0-13)
Arm/Group | Skin Adhesive | Skin Adhesive Plus Polyester Mesh
Number analyzed (Participants) | 40 | 38
Score (0-13) | 5 [5 to 6] | 5 [5 to 6]
Statistical Analysis 1: Comparison: Skin Adhesive vs Skin Adhesive Plus Polyester Mesh; Test type: Superiority; p = 0.421, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0, 95% CI 2-sided [-1 to 1], Standard Deviation 0.5

ADVERSE EVENTS:
Time Frame: From 2 weeks to 12 weeks
Arm/Group | Skin Adhesive | Skin Adhesive Plus Polyester Mesh
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 1/40 | 4/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Skin Adhesive (N=40) | Skin Adhesive Plus Polyester Mesh (N=38)
Allergic contact dermatitis (Surgical and medical procedures) | 1 (1) | 4 (4) — Mild erythema and itching at wound area, resolved with topical treatment.

LIMITATIONS AND CAVEATS:
This study has several limitations. First, it is a single-center design, so it may restrict the generalizability of our findings to other institutions and patient populations Second, all procedures were done by one experienced hip and knee arthroplasty surgeon, who had an individual technique that could have influenced wound closure quality Third, our primary outcome was the Patient and Observer which relies on patient and research assessor and may have some bias

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT06232018/Prot_SAP_000.pdf